CLINICAL TRIAL: NCT07240324
Title: The Effect of LymphaTouch® and Manual Lymphatic Drainage on Extremity Circumference Measurements in Lymphedema: A Retrospective Study
Brief Title: The Effect of LymphaTouch® and Manual Lymphatic Drainage on Extremity Circumference Measurements in Lymphedema
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: istftreah2
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MLD group: Patients with lympedema who received MLD treatment
  Interventions: Other: No intervention
- Lymphatouch group: Patients with lympedema who received Lymphatouch treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This retrospective study will be conducted using the medical records of lymphedema patients followed in the Physical Medicine and Rehabilitation outpatient clinics and lymphedema unit of Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. Women and men aged 18-75 years with a diagnosis of upper or lower extremity lymphedema will be included. Sociodemographic and clinical data of the patients will be recorded, and participants will be divided into two treatment groups: those who received LymphaTouch® therapy and those who underwent Manual Lymphatic Drainage (MLD). Pre- and post-treatment extremity circumference measurements will be obtained from patient records, and the differences between the groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with lymphedema
* Aged between 18 and 75 years
* Complete pre- and post-treatment extremity circumference measurements available in patient records

Exclusion Criteria:

* History of systemic diseases such as diabetes, rheumatologic disorders, or malignancy
* Presence of neurological disorders (e.g., polyneuropathy, multiple sclerosis, history of stroke)
* Pregnancy
* History of surgery or major trauma involving the affected limb within the past 6 months
* History of injection therapy or physical therapy applied to the same limb within the past 6 months
* History of infection or active dermatological disease affecting the limb
* Incomplete or inconsistent data in patient records

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ChatGPT:
  The study population consists of patients with lymphedema who received either LymphaTouch® or Manual Lymphatic Drainage (MLD) treatment.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Extremity Circumference (cm): | Baseline
  he primary outcome will be the difference in limb circumference measurements before and after treatment. Circumference values will be obtained from standardized anatomical landmarks, including the wrist/ankle, and at 10 cm, 20 cm, 30 cm, and 40 cm proximal to the metatarsophalangeal (MTP) or metacarpophalangeal (MCP) joint. A greater reduction in circumference indicates a more effective treatment response.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No